CLINICAL TRIAL: NCT07031622
Title: Determining the Effect of Yoga Exercises on Psychological Health and Childbirth Trauma in Pregnant Women
Brief Title: The Effect of Yoga on Mental Health and Trauma in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Collaborators: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, GÜLESER ADA, Dr, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BARU-EBE-GA-03
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2023-11

CONDITIONS: Yoga Exercises
Keywords: Childbirth trauma; pregnancy; yoga; midwife; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: In addition, preliminary information was shared with all potential participants at the beginning of the interviews were given detailed information about the research, and informed consent forms were signed. The control and intervention groups received birth preparation training for 45 minutes one day a week for 5 weeks. The experimental group additionally received a total of 10 sessions of a yoga program for 45 minutes, 2 days a week. The content of each yoga session included 10 minutes of mindful breathing, 20 minutes of yoga asanas, and 15 minutes of meditation. No yoga program was applied to the control group, and psychological assessments were not conducted. tests were performed during the same period as the experimental group. The research data for the experimental and control groups were collected from pregnant women who met the inclusion/exclusion criteria.
Masking Description: In this study, after the participants agreed to participate, they were assigned to the intervention and control groups using the simple randomization method. In the randomization process, participants were assigned odd and even numbers according to the order of application to the center. Those given odd numbers formed the intervention group. In contrast, those given even numbers formed the control group. This method was used to ensure equal distribution of the groups and to prevent selection bias. In the blinding process, the study was conducted with a single-blind design. Participants knew which group they were in, but the researchers who implemented the intervention and the statistical expert who analyzed the data were unaware of the groups' distribution, except for the person who performed the randomization. Thus, observer bias and assessment bias were minimized during the statistical analysis phase.
  This method was preferred to prevent factors that may affect participation in the i
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group additionally received a total of 10 sessions of a yoga program for 45 minutes, 2 days a week. The content of each yoga session included 10 minutes of mindful breathing, 20 minutes of yoga asanas, and 15 minutes of meditation.
  Interventions: Other: Yoga Exercises
- control (No Intervention): No intervention will be made to the control group. Only measurements will be made on parallel dates with the experimental group.

INTERVENTIONS:
Other: Yoga Exercises — The control and intervention groups received birth preparation training for 45 minutes one day a week for 5 weeks. The experimental group additionally received a total of 10 sessions of a yoga program for 45 minutes, 2 days a week. The content of each yoga session included 10 minutes of mindful breathing, 20 minutes of yoga asanas, and 15 minutes of meditation.
  Arms: Experimental group

SUMMARY:
This study aims to investigate the effects of prenatal yoga exercises on psychological health and the perception of traumatic birth in pregnant women. The study will evaluate whether a structured yoga program can reduce anxiety, improve psychological resilience, and decrease the perception of birth-related trauma during pregnancy and postpartum periods.

Study Design:

A pre-post test matched group model will be used to investigate the effects of yoga exercises. The study includes an intervention group receiving prenatal yoga training in addition to standard birth preparation education, and a control group receiving only the birth preparation education.

Population and Sample:

The study will be conducted with pregnant women applying to the obstetrics outpatient clinic of a women's and children's hospital. Eligible participants will be over 18 years of age, over 16 weeks pregnant, have a planned pregnancy, and no diagnosis of high-risk pregnancy. Exclusion criteria include hypertension, gestational diabetes, short cervical length, and low-lying placenta.

A power analysis (Type I error of 0.05, Type II error of 0.20, effect size = 0.80) determined the required sample size as 26 per group, increased to 62 in total to account for potential dropouts.

DETAILED DESCRIPTION:
Title: The Effect of Yoga on Mental Health and Trauma in Pregnant Women

Study Description (Brief Summary):

This study aims to investigate the effects of prenatal yoga exercises on psychological health and the perception of traumatic birth in pregnant women. The study will evaluate whether a structured yoga program can reduce anxiety, improve psychological resilience, and decrease the perception of birth-related trauma during pregnancy and postpartum periods.

Study Design:

A pre-post test matched group model will be used to investigate the effects of yoga exercises. The study includes an intervention group receiving prenatal yoga training in addition to standard birth preparation education, and a control group receiving only the birth preparation education.

Population and Sample:

The study will be conducted with pregnant women applying to the obstetrics outpatient clinic of a women's and children's hospital. Eligible participants will be over 18 years of age, over 16 weeks pregnant, have a planned pregnancy, and no diagnosis of high-risk pregnancy. Exclusion criteria include hypertension, gestational diabetes, short cervical length, and low-lying placenta.

A power analysis (Type I error of 0.05, Type II error of 0.20, effect size = 0.80) determined the required sample size as 26 per group, increased to 62 in total to account for potential dropouts.

Intervention:

The intervention group will attend a 5-week prenatal yoga program comprising 10 sessions (2 sessions/week, 45 minutes/session). Each session includes mindful breathing, yoga asanas, and meditation. Both groups will receive the same standard birth preparation education.

Randomization and Blinding:

Participants will be randomly assigned to intervention and control groups using simple randomization. The study is single-blind: participants will know their group, but intervention implementers and data analysts will be blinded.

Outcome Measures:

Data will be collected using the following tools:

Participant Information Form (demographic and obstetric characteristics)

Brief Psychological Resilience Scale (BPSR)

Traumatic Childbirth Perception Scale (TCPS)

Childbirth Trauma Index Scale (CTIS)

Post-Traumatic Stress Scale - Short Version

State-Trait Anxiety Inventory (STAI)

These scales will be administered pre-intervention, post-intervention, and at 7 and 40 days postpartum.

Data Analysis Plan:

Data will be analyzed using SPSS. Descriptive statistics will summarize demographic and clinical variables. Paired and independent t-tests will compare within and between-group differences. Repeated measures ANOVA will be used to assess changes in trauma perception and anxiety over time. A significance level of p<0.05 will be applied.

Ethical Considerations:

The study will be conducted following ethical principles. Ethical approval has been or will be obtained from the relevant Institutional Review Board (IRB), and informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Over 16 weeks
* Without a diagnosis of high-risk pregnancy
* Not exercising before pregnancy
* Planned pregnancy

Exclusion Criteria:

* Hypertension
* Gestational diabetes
* Short cervical length
* Low-lying placenta

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
pre-test post-test | 1 year
  This study was conducted using the "pre-post test matched group model" to investigate the effects of yoga exercises on the reduction or prevention of childbirth trauma.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No